CLINICAL TRIAL: NCT06352580
Title: Parents' Approach to Dental Treatment of Their Children in the Presence of Covid-19 Infection and Vaccine: A Pediatric Perspective
Brief Title: Covid-19 Pandemic and Pediatric Dentistry
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Deniz Sila ÖZDEMİR CELİK, assistant professor, Abant Izzet Baysal University
Other Study IDs: COVID-19 Pediatric
Record Dates: First submitted 2024-04-05; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: COVID-19 Pandemic
Keywords: Covid-19 Pandemic; Covid-19 Vaccine; Pediatric dental treatments; Dentist visit
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: It was aimed for the parents of pediatric patients to fill out the survey consisting of 26 questions. The questions were about the Covid-19 Pandemic, Covid-19 vaccines and their approach to their children's dental treatment during the Covid-19 Pandemic.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — 26 survey questions were administered face to face to parents, which they could answer in a short time.

SUMMARY:
Coronavirus (SARS-CoV-2), which emerged in Wuhan, China in 2019 and causes severe respiratory infection, poses a potential risk for dentists and patients during dental treatments. It is a common situation during the pandemic period for parents of children needing dental treatment to want to postpone their children's treatment due to Covid-19. This study aimed to evaluate parents' concerns about their children's dentist appointments and ongoing dental treatments in the presence of the quarantine imposed due to Covid-19 and the Covid-19 vaccines that have started to be administered worldwide. In the study, an informative survey consisting of 26 questions was applied to determine how parents feel about the COVID-19 pandemic, how concerned they are about their children's oral health and dental treatment plan, and the changes caused by COVID-19 vaccination practices. The questions were created by 3 different experienced dentists and analysed by 2 different experienced dentists. Questions 7 and 26 were repeated at the beginning and end of the survey to give the same question and answer meaning. Thus, the reliability of the survey was tested.

DETAILED DESCRIPTION:
This study was carried out on the parents of pediatric patients who applied to Bolu Abant İzzet Baysal University Faculty of Dentistry, Department of Pediatric Dentistry between 2022 March and 2022 June. Ethical approval of the study was approved by Bolu Abant İzzet Baysal University Clinical Research Ethics Committee (Ethics Number 2022/12). In the study, an informative survey consisting of 26 questions was applied to determine how parents feel about the COVID-19 pandemic, how concerned they are about their children's oral health and dental treatment plan, and the changes caused by COVID-19 vaccination practices (Table 1). It was aimed to apply a survey to all parents of patients who fulfilled the inclusion criteria after ethics committee approval was obtained, provided that at least 400 participants were provided.

Inclusion Criteria Being over 18 years old Volunteering for the study Being mentally healthy Parents who apply to the paediatric dentistry clinic for the treatment of their child aged 0-14 years Being able to read and understand Turkish Being a citizen of the Republic of Turkey Exclusion Criteria The patient is not accompanied by a parent Not being able to read and understand Turkish Not volunteering for the study The questions were created by 3 different experienced dentists and analysed by 2 different experienced dentists. Participants were asked questions such as their age, gender, city of residence, whether they had symptoms related to COVID-19, whether they had received dental treatment, and whether they had been vaccinated against COVID-19, and if so, which vaccine they preferred and why. In terms of the reliability of the comprehensibility of the survey, Questions 7 and 26 were repeated at the beginning and end of the survey to give the same question and answer meaning. Thus, the reliability of the survey was tested.

Statistical Analysis In this study, the relationships between categorical data were analysed by Pearson's Chi-squared Test when the sample size assumption was met (n<5) and by Fisher's Exact test when it was not met. Multiple Chi-Square test was used to investigate the relationship between multiple-choice questions. Analyses were performed in IBM SPSS 25 programme. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Volunteering for the study
* Being mentally healthy
* Parents who apply to the paediatric dentistry clinic for the treatment of their child aged 0-14 years
* Being able to read and understand Turkish
* Being a citizen of the Republic of Turkey

Exclusion Criteria:

* The patient is not accompanied by a parent
* Not being able to read and understand Turkish
* Not volunteering for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The families of the patients who came to the pediatric dentistry clinic were randomly selected from those who met the study criteria.
Sampling Method: Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Approach to dental treatments | 3 months
  How did parents approach their children's dental treatment needs in the presence of the Covid-19 pandemic?

CONTACTS AND LOCATIONS:
Locations (1):
- Deniz Sıla Özdemir Çelik, Merkez, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided